CLINICAL TRIAL: NCT03216031
Title: Project GROW: Establishing and Testing a New Intergenerational Falls Prevention Gardening Programme to Improve Physical Activity Levels, Health and Wellbeing in Older People at Risk of Falling
Brief Title: Project Grow: Establishing an Intergenerational Falls Prevention Gardening Programme
Acronym: PGROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Collaborators: St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sandra Klaperski, Senior Lecturer in Sport and Exercise Psychology, University of Roehampton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LSC/2016/55; 220793 (Other: HRA)
Record Dates: First submitted 2017-04-26; First posted 2017-07-12 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Fall
Keywords: Falls prevention; Gardening

STUDY DESIGN:
Intervention Model Description: In the implementation phase, a falls prevention gardening group will be implemented. Staff members of the Integrated Falls and Bone Health Service will offer their patients who decline to take part in the standard prevention exercise programme or who have completed the other prevention classes to participate in a gardening programme. The goal is to recruit 30 patients as participants of the gardening programme and to engage them in weekly gardening activities for 8 weeks (either 8 weeks in a row or 8 attendances over 3 months to allow for sickness / other reasons for non-attendance). 3 groups with up to 10 patients and 2-4 students/staff members each should meet once per week for about 1 hour to engage in gardening activities at the new growing site. Only participants who have passed the risk screening of the Integrated Falls and Bone Health Service and who meet all inclusion criteria will be invited to join the gardening programme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Gardening programme — 3 groups with up to 10 patients and 2-4 students/staff members each should meet once per week for about 1 hour to engage in gardening activities at the falls prevention growing site. Each participant will attend the programme 8 times.

SUMMARY:
Wandsworth Integrated Falls and Bone Health Service (IF & BHS) provides an evidence-based falls prevention exercise programme, but yearly about 500 of 1800 patients decline participation or do not continue to exercise. Our study seeks to address this efficiency gap by developing a gardening programme as an alternative to traditional exercise. In a preparation period (4/17-5/17) we will explore the special needs of the target population through interviews and create an age appropriate gardening site at "Growhampton", a gardening project run by the University of Roehampton; from 5/17 to 9/17 a falls prevention gardening group will be implemented and evaluated.

DETAILED DESCRIPTION:
The key purpose of the study is to provide and test an intergenerational gardening project as a choice for about 30 IF & BHS patients who would otherwise decline exercise interventions. Patients previously assessed by Wandsworth Integrated Falls & Bone Health Services have identified gardening as an enjoyable alternative to exercise classes. Gardening sessions will take place weekly (aiming for 3 groups with 10 patients and 2-4 students and/or staff members of the University of Roehampton). Through engaging patients in gardening activities the study seeks to achieve 4 main aims: 1. Increase physical activity levels; 2. improve mental and physical health outcomes; 3. foster self-efficacy and social connectedness; 4. reduce the risk of falls. The at falls risk population will benefit by engaging in a meaningful activity (designed and supported by clinicians and aided by students and staff members) which delivers on the core principles of strength, power, balance and coordination.

ELIGIBILITY:
Inclusion Criteria:

* Having had a Falls and Bone Health Assessment by the Integrated Falls and Bone Health Service (IF & BHS) Wandsworth
* Having falls or bone health risk factors but being able to mobilise without walking aids
* Having been assessed by IF & BHS as having capacity to take part in a gardening intervention programme
* Having indicated an interest in attending a gardening group following the IF & BHS assessment if they a) do not want to participate in any other elements of the IF & BHS programme or if they b) have completed other elements of the service offered by the IF & BHS, e.g. exercise groups, Nordic walking or Zumba gold.

Exclusion Criteria:

* Having a known diagnosis of dementia
* Not being able to adequately understand verbal explanations or written information given in English
* Having a falls risk profile that indicates that the individual has high falls risk in this context - this is a clinical decision and will take account of a number of variables including mobility (Timed up & Go of more than 20 sec) and their general health (e.g., large postural drop, uncontrolled diabetes, significant behaviour that challenges).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Physical effects 1/3 | Change in sec needed from week 1 (beginning of programme) to week 8 (end of programme)
  Timed Up and Go time (in sec)
Physical effects 2/3 | Change in number of stands achieved from week 1 (beginning of programme) to week 8 (end of programme)
  Number stands in 30 sec Sit-to-Stand test
Physical effects 3/3 | Change in numbers of steps needed from week 1 (beginning of programme) to week 8 (end of programme)
  Turn test (n steps to turn 180 degrees)
Health | Change in score achieved from week 1 (beginning of programme) to week 8 (end of programme)
  Health (EQ-5D-5L Questionnaire)
Wellbeing | Change in score achieved from week 1 (beginning of programme) to week 8 (end of programme)
  Wellbeing (Warwick-Edinburgh Mental
Falls efficacy | Change in score achieved from week 1 (beginning of programme) to week 8 (end of programme)
  Falls efficacy scale

SECONDARY OUTCOMES:
Falls and incidents | Number of falls/incidents recorded during the programme (week 1-8)
  Number of falls or other incidences during the gardening programme to judge its feasibility and risks.
Activity levels | Change from week 1 (beginning of programme) to week 8 (end of programme)
  Activity Levels (assessed by means of interview question)
Self-efficacy | Change in score achieved from week 1 (beginning of programme) to week 8 (end of programme)
  General self-efficacy scale
Social connectedness | Change in score achieved from week 1 (beginning of programme) to week 8 (end of programme)
  Social connectedness scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Roehampton in collaboration with St George's University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No